CLINICAL TRIAL: NCT00447876
Title: Double-blind, Placebo-controlled, Randomised, Multicentre Study on the Efficacy and Safety of a Single Injection of Botulinum Toxin A (200 Units Dysport®) in the Treatment of Chronic Plantar Fasciitis
Brief Title: Study to Assess the Efficacy and Safety of Dysport® in the Treatment of Chronic Plantar Fasciitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-94-52120-100; 2004-002533-39 (EudraCT Number)
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Chronic Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum type A toxin (Dysport®) (Experimental)
  Interventions: Biological: Botulinum toxin type A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — Botulinum type A toxin (Dysport®): 200 Units injected at the root of the plantar fascia
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Botulinum type A toxin (Dysport®)
Drug: Placebo — 0.9% sodium chloride: 2 ml injected at the root of the plantar fascia
  Arms: Placebo

SUMMARY:
This study will investigate the hypothesis that the analgesic effect of a single injection of Dysport (200 MU) induces a significant reduction of symptoms in chronic cases of plantar fasciitis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plantar fasciitis (duration of disorder at least 4 months)
* At least 4 points on the visual analogue scale (0-10) for the most severe pain within the last 48 hours
* At least 2 previous unsuccessful conservative therapies
* Age 18 and older

Exclusion Criteria:

* Rheumatoid diseases (M. Bechterew, chronic polyarthritis, psoriasis-arthritis, para /post-infectious arthritis etc.)
* Previous surgery in the affected area of the foot
* Pre-treatment with Botulinum toxin A (only de novo patients)
* Prohibited concomitant treatment: local injections during the study and 2 weeks prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-07; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (6):
- Germany (6):
  - University Hospital Charite, Campus Virchow, Musculoskeletal Centre, Orthopedic Clinic, Berlin
  - Orthopedic Practice Biberburg, Berlin
  - Orthopedic Practice, Karlsruhe
  - Klinik für Orthopädie und Rheumatologie, Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Orthocentre Munich, Munich
  - Orthopedic Practice, Weiden

REFERENCES:
- [Result] Peterlein CD, Funk JF, Holscher A, Schuh A, Placzek R. Is botulinum toxin A effective for the treatment of plantar fasciitis? Clin J Pain. 2012 Jul;28(6):527-33. doi: 10.1097/AJP.0b013e31823ae65a. PMID 22673486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a double-blind, placebo-controlled, randomized, prospective study where patients were recruited to 5 study centres in Germany. Patients were enrolled to the study from 08 July 2005 (first patent enrolled) until 23 April 2009 (last patient completed).
Pre-assignment Details: 40 patients were enrolled. Patients were assigned to treatment if they met all inclusion and none of the exclusion criteria. All patients enrolled were randomized and received study treatment.
Groups:
- Dysport ® 200 U: Patients received one injection of 200 units (U) Dysport® at Week 0 (Day 0). The study treatment was injected into the origin of the plantar fascia in accordance with the clinical findings on palpation, the injection being distributed in four portions in a fan-shaped manner using a single 0.50 x 40mm needle. Follow-up examinations to assess the efficacy and safety of the treatment were performed at Weeks 2, 6, 10, 14 and 18.
- Placebo: Patients received one injection of placebo (physiological sodium chloride solution, 2ml) at Week 0 (Day 0). The study treatment was injected into the origin of the plantar fascia in accordance with the clinical findings on palpation, the injection being distributed in four portions in a fan-shaped manner using a single 0.50 x 40mm needle. Follow-up examinations to assess the efficacy and safety of the treatment were performed at Weeks 2, 6, 10, 14 and 18.
Period: Overall Study
Arm/Group | Dysport ® 200 U | Placebo
Started | 20 | 20
Completed | 17 | 16
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Deterioration of symptomology | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for all patients randomized in the study.
Arm/Group | Dysport ® 200 U | Placebo | Total Title
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.7) | 51.8 (11.3) | 52.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 32
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Responders Rate at Week 6 (Pain While Moving)
Description: The responder rate was defined as the percentage of patients whose pain score while moving during the last 48 hours, measured by means of a 10 cm Visual Analogue Scale (VAS, 0 = no pain, 10 = maximum pain) decreased by at least 50% at Week 6 as compared to baseline. Pain at movement is the cardinal symptom of plantar fasciitis and the 10 cm VAS is a reference method for the assessment of pain intensity.
Time Frame: Baseline and Week 6
Population: The Intention-To-Treat (ITT) analysis set was defined as the set of randomized patients who received study treatment and for whom values of the efficacy parameters were available at baseline and at least once at a later timepoint. Missing values were replaced using the last observation carried forward (LOCF) method.
Measure: Number; unit: Percentage of participants
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
Percentage of participants | 25.0 | 5.0
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; The responders rate at Week 6 was compared between treatment groups by a two-sided Fisher exact test; Test type: Superiority or Other; p = 0.182, Fisher Exact; Treatment difference = 0.20, 95% CI 2-sided [-0.06 to 0.46]

2. Secondary Outcome: Changes From Baseline in Gerbershagen's Score at Week 18
Description: The Gerbershagen scale gives a global score ranging between I and III, with lower scores reflecting less impact of pain in terms of temporal, spatial aspects, drug taking behaviour and utilization of the health care system. The changes in Gerbershagen's global scores from baseline to Week 18 are reported as percentage of patients for each of the specified categories.
Time Frame: Baseline and Week 18
Population: The ITT analysis set was defined as the set of randomized patients who received study treatment and for whom values of the efficacy parameters were available at baseline and at least one later timepoint. This variable could only be analyzed for 30 patients (15 from each group) for whom the score could be determined both at baseline and at Week 18.
Measure: Number; unit: Percentage of participants
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 15 | 15
Percentage of participants
  Baseline score = I; Week 18 score = I | 40.0 | 60.0
  Baseline score = II; Week 18 score = I | 26.7 | 6.7
  Baseline score = II; Week 18 score = II | 6.7 | 20.0
  Baseline score = II; Week 18 score = III | 6.7 | 0.0
  Baseline score = III; Week 18 score = I | 6.7 | 6.7
  Baseline score = III; Week 18 score = II | 6.7 | 6.7
  Baseline score = III; Week 18 score = III | 6.7 | 0.0
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; Gerbershagen's Global scores were compared at Week 18 using a Cochran-Mantel-Haenszel analysis of variance statistic with adjustment to the baseline score; Test type: Superiority or Other; p = 0.222, Cochran-Mantel-Haenszel

3. Secondary Outcome: Changes From Baseline in Maximum Pain (Pain While Moving) at Each Visit
Description: Assessments of the pain intensity while moving (maximum pain during the previous 48 hours) were performed by means of a 10 cm VAS (0 = no pain, 10 = maximum pain) at each visit. The changes from baseline, expressed as Pain Intensity Difference (PID) values at each indicated timepoint are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: The ITT analysis set was defined as the set of randomized patients who received study treatment and for whom values of the efficacy parameters were available at baseline and at least one later timepoint. Missing values were replaced using the LOCF method.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
Centimeter (cm)
  PID Week 2 (maximum pain) | -1.38 (2.66) | -1.18 (1.98)
  PID Week 6 (maximum pain) | -1.55 (3.27) | -1.35 (1.85)
  PID Week 10 (maximum pain) | -1.75 (3.32) | -1.25 (1.99)
  PID Week 14 (maximum pain) | -2.48 (3.59) | -1.30 (2.59)
  PID Week 18 (maximum pain) | -2.45 (3.52) | -1.80 (3.17)

4. Secondary Outcome: Assessment of Sum of Pain Intensity Difference (SPID) for Maximum Pain for Overall Study
Description: Assessments of the pain intensity while moving (maximum pain during the previous 48 hours) were performed by means of a 10 cm VAS (0 = no pain, 10 = maximum pain) at each visit. The PID values at each timepoint were determined by comparison to baseline, followed by calculation of the area under the curve (AUC) of PID as a function of time (i.e. SPID). The least square (LS) means of SPID, adjusted for the baseline value of pain while moving are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: cm * day
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
cm * day | -28.043 [-43.672 to -12.415] | -19.207 [-34.835 to -3.578]
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; SPID was compared between the two treatment groups using a fixed effect analysis of covariance (ANCOVA) taking into account the SPID value as dependent variable, the baseline pain intensity as co-variable, and the treatment group as explicative variable; Test type: Superiority or Other; p = 0.423, ANCOVA; LS mean difference = -8.837, 95% CI 2-sided [-30.940 to 13.266]

5. Secondary Outcome: Changes From Baseline in Continuous Pain (Pain At Rest) at Each Visit
Description: Assessments of the pain intensity while at rest (continuous pain during the previous 48 hours) were performed by means of a 10 cm VAS (0 = no pain, 10 = maximum pain) at each visit. The changes from baseline, expressed as PID values at each indicated timepoint are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
cm
  PID Week 2 (continuous pain) | -0.78 (2.80) | -0.88 (2.19)
  PID Week 6 (continuous pain) | -0.45 (2.70) | -1.05 (1.76)
  PID Week 10 (continuous pain) | -0.63 (2.67) | -1.20 (2.98)
  PID Week 14 (continuous pain) | -1.75 (2.99) | -0.98 (2.91)
  PID Week 18 (continuous pain) | -1.55 (3.38) | -1.70 (3.75)

6. Secondary Outcome: Assessment of SPID for Continuous Pain for Overall Study
Description: Assessments of the pain intensity while at rest (continuous pain during the previous 48 hours) were performed by means of a 10 cm VAS (0 = no pain, 10 = maximum pain) at each visit. The PID values at each timepoint were determined by comparison to baseline, followed by calculation of the AUC of PID as a function of time (i.e. SPID). The LS means for SPID, adjusted for the baseline value of pain at rest are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: cm * day
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
cm * day | -17.511 [-31.838 to -3.184] | -13.339 [-27.666 to 0.988]
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; SPID was compared between the two treatment groups using a fixed effect ANCOVA taking into account the SPID value as dependent variable, the baseline pain intensity as co-variable, and the treatment group as explicative variable; Test type: Superiority or Other; p = 0.682, ANCOVA; LS mean difference = -4.173, 95% CI 2-sided [-24.640 to 16.294]

7. Secondary Outcome: Changes From Baseline in Pain Threshold at Each Visit
Description: The maximum pain felt in the medial back foot was measured using an algometer. The pain threshold corresponded to the maximum pressure at which pain was still tolerated. Changes from baseline, expressed as pain threshold differences at each indicated timepoint are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Kilogram (kg) / cm^2
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
Kilogram (kg) / cm^2
  Pain threshold difference Week 2 | 0.80 (2.28) | 0.76 (1.73)
  Pain threshold difference Week 6 | 0.51 (2.90) | 1.31 (3.95)
  Pain threshold difference Week 10 | 0.69 (2.86) | 1.50 (3.51)
  Pain threshold difference Week 14 | 0.85 (3.41) | 1.35 (2.97)
  Pain threshold difference Week 18 | 0.83 (3.23) | 2.16 (3.93)

8. Secondary Outcome: Assessment of Sum of Pain Threshold Differences (by Measurement of AUC) for Overall Study
Description: Assessments of the pain threshold using an algometer (which was the pressure corresponding to the maximum tolerated pain) were performed at each visit. Pain threshold differences at each timepoint were determined by comparison to baseline, followed by calculation of the AUC of the pain threshold difference as a function of time. The LS means of AUC, adjusted for the baseline value of pain threshold are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: (kg / cm^2) * day
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
(kg / cm^2) * day | 11.492 [-3.238 to 26.223] | 19.558 [4.827 to 34.288]
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; The sum of pain threshold difference (i.e. SPID expressed as AUC) was compared between the two treatment groups using a fixed effect ANCOVA taking into account the SPID AUC value as dependent variable, the baseline pain intensity as co-variable, and the treatment group as explicative variable; Test type: Superiority or Other; p = 0.438, ANCOVA; LS mean difference = -8.066, 95% CI 2-sided [-28.910 to 12.779]

9. Secondary Outcome: Changes From Baseline in Pressure Threshold (With Algometer) at Each Visit
Description: Pressure pain in the medial back foot was measured using an algometer. Pressure threshold corresponded to the minimum pressure causing pain. The changes from baseline, expressed as pressure threshold differences at each indicated timepoint are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg / cm^2
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
kg / cm^2
  Pressure threshold difference Week 2 | 0.55 (2.21) | 0.95 (1.76)
  Pressure threshold difference Week 6 | 0.90 (2.62) | 1.07 (2.01)
  Pressure threshold difference Week 10 | 0.61 (1.79) | 1.33 (2.29)
  Pressure threshold difference Week 14 | 1.38 (2.77) | 1.13 (2.20)
  Pressure threshold difference Week 18 | 1.74 (2.98) | 1.28 (2.47)

10. Secondary Outcome: Assessment of Sum of Pressure Threshold Differences (by Measurement of AUC) for Overall Study
Description: Assessments of the pressure threshold using an algometer (which corresponded to the minimum pressure causing pain) were performed at each visit. Pressure threshold differences at each timepoint were determined by comparison to baseline, followed by calculation of the AUC of the pressure threshold difference as a function of time. The LS means of AUC, adjusted for the baseline value of pressure threshold are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: (kg / cm^2) * day
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
(kg / cm^2) * day | 16.174 [5.462 to 26.886] | 15.581 [4.869 to 26.293]
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; The sum of pressure threshold difference (i.e. SPID expressed as AUC) was compared between the two treatment groups using a fixed effect ANCOVA taking into account the SPID AUC value as dependent variable, the baseline pain intensity as co-variable, and the treatment group as explicative variable; Test type: Superiority or Other; p = 0.937, ANCOVA; LS mean difference = 0.594, 95% CI 2-sided [-14.575 to 15.762]

11. Secondary Outcome: Assessment of Dorsal Extension / Plantar Flexion Range of Motion (ROM) of the Affected Foot At Week 18
Description: Dorsal extension and plantar flexion of the affected foot were assessed at baseline and at Week 18. A ROM of approximately 70 degrees is considered to be normal. The LS means, adjusted for the baseline value are reported.
Time Frame: Baseline and Week 18
Population: The ITT analysis set was defined as the set of randomized patients who received study treatment and for whom values of the efficacy parameters were available at baseline and at least one later timepoint. This variable was only analyzed for 34 patients (18 for Dysport® and 16 for Placebo) for whom ROM was determined at both baseline and Week 18.
Measure: Least Squares Mean (95% Confidence Interval); unit: Degrees
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 18 | 16
Degrees | 60.7 [56.6 to 64.8] | 61.4 [57.1 to 65.8]
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; Test type: Superiority or Other; p = 0.800, ANCOVA — The difference (most affected side - control side) in ROM for the dorsal extension was analyzed using a fixed effect ANCOVA, using Week 18 results as the dependent variable and baseline value as covariate; LS mean difference = -0.8, 95% CI 2-sided [-6.8 to 5.3]

12. Secondary Outcome: Number of Patients Without Pain and/or With a Pain Reduction Based on Global Assessment of Pain by Investigator at Each Visit
Description: A global assessment of the patient's current condition relative to baseline was performed by the Investigator at each visit using 5 level scale: significantly better, slightly better, unchanged, slightly worse, significantly worse. The number of patients for each variable at each indicated timepoint are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: The ITT analysis set was defined as the set of randomized patients who received study treatment and for whom values of the efficacy parameters were available at baseline and at least one later timepoint.
Measure: Number; unit: Number of participants
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
Number of participants
  Week 2 significantly worse: number analyzed (Participants) | 20 | 18
  Week 2 significantly worse | 0 | 0
  Week 2 slightly worse: number analyzed (Participants) | 20 | 18
  Week 2 slightly worse | 1 | 0
  Week 2 unchanged: number analyzed (Participants) | 20 | 18
  Week 2 unchanged | 9 | 9
  Week 2 slightly improved: number analyzed (Participants) | 20 | 18
  Week 2 slightly improved | 7 | 6
  Week 2 significantly improved: number analyzed (Participants) | 20 | 18
  Week 2 significantly improved | 3 | 3
  Week 6 significantly worse: number analyzed (Participants) | 19 | 20
  Week 6 significantly worse | 2 | 2
  Week 6 slightly worse: number analyzed (Participants) | 19 | 20
  Week 6 slightly worse | 0 | 0
  Week 6 unchanged: number analyzed (Participants) | 19 | 20
  Week 6 unchanged | 6 | 9
  Week 6 slightly improved: number analyzed (Participants) | 19 | 20
  Week 6 slightly improved | 7 | 8
  Week 6 significantly improved: number analyzed (Participants) | 19 | 20
  Week 6 significantly improved | 4 | 1
  Week 10 significantly worse: number analyzed (Participants) | 16 | 19
  Week 10 significantly worse | 2 | 3
  Week 10 slightly worse: number analyzed (Participants) | 16 | 19
  Week 10 slightly worse | 2 | 2
  Week 10 unchanged: number analyzed (Participants) | 16 | 19
  Week 10 unchanged | 2 | 3
  Week 10 slightly improved: number analyzed (Participants) | 16 | 19
  Week 10 slightly improved | 7 | 10
  Week 10 significantly improved: number analyzed (Participants) | 16 | 19
  Week 10 significantly improved | 3 | 1
  Week 14 significantly worse: number analyzed (Participants) | 18 | 17
  Week 14 significantly worse | 2 | 1
  Week 14 slightly worse: number analyzed (Participants) | 18 | 17
  Week 14 slightly worse | 1 | 1
  Week 14 unchanged: number analyzed (Participants) | 18 | 17
  Week 14 unchanged | 4 | 5
  Week 14 slightly improved: number analyzed (Participants) | 18 | 17
  Week 14 slightly improved | 7 | 7
  Week 14 significantly improved: number analyzed (Participants) | 18 | 17
  Week 14 significantly improved | 4 | 3
  Week 18 significantly worse: number analyzed (Participants) | 18 | 20
  Week 18 significantly worse | 2 | 5
  Week 18 slightly worse: number analyzed (Participants) | 18 | 20
  Week 18 slightly worse | 0 | 0
  Week 18 unchanged: number analyzed (Participants) | 18 | 20
  Week 18 unchanged | 4 | 3
  Week 18 slightly improved: number analyzed (Participants) | 18 | 20
  Week 18 slightly improved | 6 | 8
  Week 18 significantly improved: number analyzed (Participants) | 18 | 20
  Week 18 significantly improved | 6 | 4
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 2. The variables for global assessment of pain assessed by the Investigator were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.862, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 6. The variables for global assessment of pain assessed by the Investigator were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.317, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 10. The variables for global assessment of pain assessed by the Investigator were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.525, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 14. The variables for global assessment of pain assessed by the Investigator were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.931, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 18. The variables for global assessment of pain assessed by the Investigator were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.353, Wilcoxon rank sum test

13. Secondary Outcome: Number of Patients Without Pain and/or With a Pain Reduction Based on Global Assessment of Pain by Patient at Each Visit
Description: A global assessment of the patient's current condition relative to baseline was performed by the patient at each visit using a 5 level scale: significantly better, slightly better, unchanged, slightly worse, significantly worse. The number of patients for each variable at each indicated timepoint are reported.
Time Frame: Baseline and Weeks 2, 6, 10, 14 and 18
Population: as for outcome 12
Measure: Number; unit: Number of participants
Arm/Group | Dysport ® 200 U | Placebo
Number analyzed (Participants) | 20 | 20
Number of participants
  Week 2 significantly worse: number analyzed (Participants) | 20 | 19
  Week 2 significantly worse | 0 | 0
  Week 2 slightly worse: number analyzed (Participants) | 20 | 19
  Week 2 slightly worse | 3 | 2
  Week 2 unchanged: number analyzed (Participants) | 20 | 19
  Week 2 unchanged | 7 | 9
  Week 2 slightly improved: number analyzed (Participants) | 20 | 19
  Week 2 slightly improved | 7 | 5
  Week 2 significantly improved: number analyzed (Participants) | 20 | 19
  Week 2 significantly improved | 3 | 3
  Week 6 significantly worse: number analyzed (Participants) | 19 | 20
  Week 6 significantly worse | 3 | 2
  Week 6 slightly worse: number analyzed (Participants) | 19 | 20
  Week 6 slightly worse | 0 | 1
  Week 6 unchanged: number analyzed (Participants) | 19 | 20
  Week 6 unchanged | 6 | 9
  Week 6 slightly improved: number analyzed (Participants) | 19 | 20
  Week 6 slightly improved | 6 | 6
  Week 6 significantly improved: number analyzed (Participants) | 19 | 20
  Week 6 significantly improved | 4 | 2
  Week 10 significantly worse: number analyzed (Participants) | 17 | 19
  Week 10 significantly worse | 4 | 3
  Week 10 slightly worse: number analyzed (Participants) | 17 | 19
  Week 10 slightly worse | 2 | 2
  Week 10 unchanged: number analyzed (Participants) | 17 | 19
  Week 10 unchanged | 3 | 3
  Week 10 slightly improved: number analyzed (Participants) | 17 | 19
  Week 10 slightly improved | 4 | 7
  Week 10 significantly improved: number analyzed (Participants) | 17 | 19
  Week 10 significantly improved | 4 | 4
  Week 14 significantly worse: number analyzed (Participants) | 18 | 17
  Week 14 significantly worse | 2 | 1
  Week 14 slightly worse: number analyzed (Participants) | 18 | 17
  Week 14 slightly worse | 3 | 2
  Week 14 unchanged: number analyzed (Participants) | 18 | 17
  Week 14 unchanged | 3 | 4
  Week 14 slightly improved: number analyzed (Participants) | 18 | 17
  Week 14 slightly improved | 7 | 5
  Week 14 significantly improved: number analyzed (Participants) | 18 | 17
  Week 14 significantly improved | 3 | 5
  Week 18 significantly worse: number analyzed (Participants) | 19 | 20
  Week 18 significantly worse | 3 | 5
  Week 18 slightly worse: number analyzed (Participants) | 19 | 20
  Week 18 slightly worse | 2 | 0
  Week 18 unchanged: number analyzed (Participants) | 19 | 20
  Week 18 unchanged | 2 | 4
  Week 18 slightly improved: number analyzed (Participants) | 19 | 20
  Week 18 slightly improved | 5 | 7
  Week 18 significantly improved: number analyzed (Participants) | 19 | 20
  Week 18 significantly improved | 7 | 4
Statistical Analysis 1: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 2. The variables for global assessment of pain assessed by the patient were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.882, Wilcoxon rank sum test
Statistical Analysis 2: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 6. The variables for global assessment of pain assessed by the patient were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.489, Wilcoxon rank sum test
Statistical Analysis 3: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 10. The variables for global assessment of pain assessed by the patient were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.660, Wilcoxon rank sum test
Statistical Analysis 4: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 14. The variables for global assessment of pain assessed by the patient were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.485, Wilcoxon rank sum test
Statistical Analysis 5: Comparison: Dysport ® 200 U vs Placebo; Dysport® vs placebo at Week 18. The variables for global assessment of pain assessed by the patient were described at each visit as ordinal qualitative variables and were compared between the two treatment groups by means of a non parametric Wilcoxon rank sum test; Test type: Superiority or Other; p = 0.392, Wilcoxon rank sum test

ADVERSE EVENTS:
Time Frame: Up to Week 18
Description: Adverse events are described in terms of incidence of Treatment Emergent Adverse Events. Safety was assessed on all randomized patients who received study treatment and were assessed for safety at least once after baseline.
Arm/Group | Dysport ® 200 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 8/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport ® 200 U (N=20) | Placebo (N=20)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport ® 200 U (N=20) | Placebo (N=20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No